CLINICAL TRIAL: NCT01610050
Title: A Phase I, Multicenter, Open-label Study of LFA102 Administered Intravenously in Japanese Patients With Castration-resistant Prostate Cancer or Advanced Breast Cancer
Brief Title: A Phase I Study of LFA102 in Japanese Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLFA102X1101
Record Dates: First submitted 2012-05-30; First posted 2012-06-01 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Castration-resistant Prostate Cancer, Advanced Breast Cancer
Keywords: castration-resistant prostate cancer, advanced breast cancer
MeSH Terms: interventions — LFA102 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LFA102 (Experimental)
  Interventions: Drug: LFA102

INTERVENTIONS:
Drug: LFA102
  Other Names: anti prolactin receptor humanized monoclonal antibody

SUMMARY:
This study will evaluate safety and tolerability to determine the MTD/RD.

DETAILED DESCRIPTION:
This is a phase I open-label, multi-center, dose escalation study in Japanese patients with CRPC or advanced BC. LFA102 will be administered intravenously once every 4 weeks during the study. All patients will remain on treatment until they meet the criteria for study discontinuation (e.g. disease progression, unacceptable toxicity, patient withdrawal) or study closure.

This study is to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of LFA102. Each cohort will enroll a minimum of 3 patients. A two-parameter Bayesian logistic regression model employing the escalation with overdose control principle will be used during the escalation phase for dose level selection and for determination of the MTD or RD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate cancer
* Histologically or cytologically confirmed locally advanced or metastatic breast cancer

Exclusion Criteria:

* Patients with untreated and/or symptomatic metastatic CNS disease
* Prior anaphylactic or other severe infusion reaction
* Treatment with agent which affect prolactin levels
* Active autoimmune disease

Other protcol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | 1st treatment cycle (28 days)
  Frequency and severity of dose limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Frequency, duration and severity of Adverse Events (AEs) | at informed consent, until 28 days after treatment discontinuation
  Frequency, duration and severity of all AEs will be collected.
Serum Concentration | cycle 1 day 1 until disease progression
Objective Response Rate | every 8 week or 12 weeks, until disase progression
  Assessed based on RECIST/PCWG2 criteria
Antibodies against LFA102 | day 1 of each treatment cycle until disease progression
  Serum concentration of antibodies against LFA102
Progression Free Survival | every 8 or 12 weeks until disease progression
  Assessed based on RECIST/PCWG2 criteria
PK parameters | cycle 1 day 1 until disease progression
  Cmax, Tmax, AUC, T1/2, CL and V

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Chuo-ku, Tokyo